CLINICAL TRIAL: NCT06201182
Title: Efficacy of Fecal Microbiota Transplantation (FMT) in Irritable Bowel Syndrome (IBS): A Randomized, Placebo-controlled, Double-blind Study
Brief Title: Efficacy of Fecal Microbiota Transplantation (FMT) in Irritable Bowel Syndrome (IBS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Natsuda Aumpan, MD, Principal Investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MTU-EC-IM-1-080/63
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: Fecal microbiota transplantation
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into 3 groups:
  * In placebo group, patients will receive placebo capsules and placebo via enema.
  * In enema group, patients will receive placebo capsules and FMT via rectal enema.
  * In capsule group, patients will receive FMT capsules and placebo via rectal enema.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FMT rectal enema (Experimental): Patients will receive FMT via rectal enema and placebo capsules.
  Interventions: Drug: FMT via rectal enema; Drug: Placebo capsules
- Encapsulated FMT (Experimental): Patients will receive FMT capsules and placebo via rectal enema.
  Interventions: Drug: FMT capsules; Drug: Placebo via rectal enema
- Placebo (Placebo Comparator): Patients will receive placebo capsules and placebo via rectal enema.
  Interventions: Drug: Placebo via rectal enema; Drug: Placebo capsules

INTERVENTIONS:
Drug: FMT via rectal enema — 50 grams of FMT via rectal enema
  Arms: FMT rectal enema
Drug: FMT capsules — FMT capsules given twice daily for 2 consecutive days
  Arms: Encapsulated FMT
Drug: Placebo via rectal enema — Placebo via rectal enema
  Arms: Encapsulated FMT; Placebo
Drug: Placebo capsules — Placebo capsules given twice daily for 2 consecutive days
  Arms: FMT rectal enema; Placebo

SUMMARY:
The goal of this clinical trial is to determine efficacy of FMT via rectal enema and encapsulated FMT in patients with IBS in Thailand. The main question it aims to answer is:

• Does FMT provide better efficacy than placebo in IBS patients?

Participants will be randomized into 3 groups:

* In placebo group, patients will receive placebo capsules and placebo via enema.
* In enema group, patients will receive placebo capsules and FMT via rectal enema.
* In capsule group, patients will receive FMT capsules and placebo via rectal enema.

Researchers will compare FMT and placebo group to see if using FMT provides better efficacy for IBS patients than placebo. Moreover, researchers will compare efficacy of FMT capsules and FMT via rectal enema in IBS patients.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a common functional bowel disorder defined by recurrent abdominal pain related to defecation or a change in bowel habit (1). Pathogenic mechanisms of IBS include gut microbial dysbiosis, low-grade mucosal inflammation, increased gut permeability, and altered gut-brain interaction (2). Dysbiosis is an imbalance of gut microbiota which can contribute to IBS. Emerging treatment approach for IBS aims to correct dysbiosis by modulation of intestinal microbiota (3).

Fecal microbiota transplantation (FMT) is an administration of feces from a healthy donor to the gastrointestinal tract of a recipient in order to restore balanced microbial flora (4). Correcting gut dysbiosis might be another target to improve IBS symptoms. Some previous randomized controlled trials demonstrated that FMT could provide clinical response in patients with IBS (5-7), whereas others reported no different outcome from placebo (8, 9). Most trials delivered FMT via more invasive routes such as colonoscopy or gastroscopy. There were few studies using less invasive methods, e.g., oral FMT capsules and FMT via rectal enema. Less invasive routes of FMT administration are needed to be evaluated so as to reduce risk and cost of endoscopy.

This study aimed to determine efficacy of FMT via rectal enema and encapsulated FMT compared with placebo in IBS patients in Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years with IBS diagnosed by Rome IV criteria
* Patients who can provide written informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Severe comorbidities: chronic kidney disease (GFR<15 ml/min), cirrhosis, cancer, etc.
* Fecal incontinence
* Immunocompromised patients
* Taking probiotic, or fermented food
* Discontinue medication for IBS <1 month prior to study inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2024-08-19 (Estimated); Study Completion 2024-08-19 (Estimated)

PRIMARY OUTCOMES:
The proportion of responders | 4 weeks, 12 weeks
  Response is defined as a decrease in IBS-symptom severity score (IBS-SSS) more than 50 points from baseline.

SECONDARY OUTCOMES:
Quality of life score | 4 weeks, 12 weeks
  Quality of life score will be assessed in both FMT and placebo groups
Adverse event | 4 weeks, 12 weeks
  Record adverse events during and after treatment
Changes in microbiota diversity before and after FMT | 4 weeks
  Evaluate changes in microbiota diversity before and after FMT

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University, Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mearin F, Lacy BE, Chang L, Chey WD, Lembo AJ, Simren M, Spiller R. Bowel Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00222-5. doi: 10.1053/j.gastro.2016.02.031. Online ahead of print. PMID 27144627
- [Background] Holtmann GJ, Ford AC, Talley NJ. Pathophysiology of irritable bowel syndrome. Lancet Gastroenterol Hepatol. 2016 Oct;1(2):133-146. doi: 10.1016/S2468-1253(16)30023-1. Epub 2016 Sep 8. PMID 28404070
- [Background] Simren M, Barbara G, Flint HJ, Spiegel BM, Spiller RC, Vanner S, Verdu EF, Whorwell PJ, Zoetendal EG; Rome Foundation Committee. Intestinal microbiota in functional bowel disorders: a Rome foundation report. Gut. 2013 Jan;62(1):159-76. doi: 10.1136/gutjnl-2012-302167. Epub 2012 Jun 22. PMID 22730468
- [Background] Cammarota G, Ianiro G, Tilg H, Rajilic-Stojanovic M, Kump P, Satokari R, Sokol H, Arkkila P, Pintus C, Hart A, Segal J, Aloi M, Masucci L, Molinaro A, Scaldaferri F, Gasbarrini G, Lopez-Sanroman A, Link A, de Groot P, de Vos WM, Hogenauer C, Malfertheiner P, Mattila E, Milosavljevic T, Nieuwdorp M, Sanguinetti M, Simren M, Gasbarrini A; European FMT Working Group. European consensus conference on faecal microbiota transplantation in clinical practice. Gut. 2017 Apr;66(4):569-580. doi: 10.1136/gutjnl-2016-313017. Epub 2017 Jan 13. PMID 28087657
- [Background] El-Salhy M, Hatlebakk JG, Gilja OH, Brathen Kristoffersen A, Hausken T. Efficacy of faecal microbiota transplantation for patients with irritable bowel syndrome in a randomised, double-blind, placebo-controlled study. Gut. 2020 May;69(5):859-867. doi: 10.1136/gutjnl-2019-319630. Epub 2019 Dec 18. PMID 31852769
- [Background] Holvoet T, Joossens M, Vazquez-Castellanos JF, Christiaens E, Heyerick L, Boelens J, Verhasselt B, van Vlierberghe H, De Vos M, Raes J, De Looze D. Fecal Microbiota Transplantation Reduces Symptoms in Some Patients With Irritable Bowel Syndrome With Predominant Abdominal Bloating: Short- and Long-term Results From a Placebo-Controlled Randomized Trial. Gastroenterology. 2021 Jan;160(1):145-157.e8. doi: 10.1053/j.gastro.2020.07.013. Epub 2020 Jul 15. PMID 32681922
- [Background] Johnsen PH, Hilpusch F, Cavanagh JP, Leikanger IS, Kolstad C, Valle PC, Goll R. Faecal microbiota transplantation versus placebo for moderate-to-severe irritable bowel syndrome: a double-blind, randomised, placebo-controlled, parallel-group, single-centre trial. Lancet Gastroenterol Hepatol. 2018 Jan;3(1):17-24. doi: 10.1016/S2468-1253(17)30338-2. Epub 2017 Nov 1. PMID 29100842
- [Background] Halkjaer SI, Christensen AH, Lo BZS, Browne PD, Gunther S, Hansen LH, Petersen AM. Faecal microbiota transplantation alters gut microbiota in patients with irritable bowel syndrome: results from a randomised, double-blind placebo-controlled study. Gut. 2018 Dec;67(12):2107-2115. doi: 10.1136/gutjnl-2018-316434. Epub 2018 Jul 6. PMID 29980607
- [Background] Aroniadis OC, Brandt LJ, Oneto C, Feuerstadt P, Sherman A, Wolkoff AW, Kassam Z, Sadovsky RG, Elliott RJ, Budree S, Kim M, Keller MJ. Faecal microbiota transplantation for diarrhoea-predominant irritable bowel syndrome: a double-blind, randomised, placebo-controlled trial. Lancet Gastroenterol Hepatol. 2019 Sep;4(9):675-685. doi: 10.1016/S2468-1253(19)30198-0. Epub 2019 Jul 17. PMID 31326345
- [Derived] Aumpan N, Chonprasertsuk S, Pornthisarn B, Siramolpiwat S, Bhanthumkomol P, Issariyakulkarn N, Gamnarai P, Bongkotvirawan P, Wongcha-Um A, Mahachai V, Vilaichone RK. Efficacy of encapsulated fecal microbiota transplantation and FMT via rectal enema for irritable bowel syndrome: a double-blind, randomized, placebo-controlled trial (CAP-ENEMA FMT Trial). Front Med (Lausanne). 2025 Sep 23;12:1648944. doi: 10.3389/fmed.2025.1648944. eCollection 2025. PMID 41064515